CLINICAL TRIAL: NCT02147782
Title: Continuous Clinical Observation on Bone Metabolism Induced by Chronic Renal Insufficiency in Different Stages
Brief Title: Clinical Observation on Bone Metabolism Induced by Chronic Renal Insufficiency
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Anhui Provincial Hospital (Other Government); Huadong Hospital (Other); Longhua Hospital (Other)
Responsible Party: Principal Investigator, Bing Shu, Associate Professor, Shanghai University of Traditional Chinese Medicine
Other Study IDs: Renal Osteodystrophy; 1RT1270,2010CB530400 (Other Grant/Funding Number: Innovative Research Team in University of Ministry of Education of China, 973 Project)
Record Dates: First submitted 2014-05-13; First posted 2014-05-28 (Estimated); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Chronic Renal Insufficiency; Renal Osteodystrophy
Keywords: chronic renal insufficient, renal osteodystrophy, bone mineral density, bone turnover, kidney function
MeSH Terms: conditions — Renal Insufficiency, Chronic; Chronic Kidney Disease-Mineral and Bone Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Serum and plasma of cases and controls
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- control: Healthy people from physical examination centers are recruited as controls.
- CKD1: 1. with clinical one or more symptoms and signs of kidney injury listed as below：
     1. Urinary albumin ( urinary albumin excretion rate≥30 mg/24 h.albumin-creatinine ratio≥3mg/mmol)
     2. urinary sediments abnormality
     3. renal tubular lesions
     4. renal histological abnormalities
     5. abnormal structure showed by imaging
     6. history of renal transplantation
  2. GFR≥90（ml/min/1.73m²)
- CKD2: with clinical symptoms and signs of kidney injury, and 60<=GFR<=89（ml/min/1.73m²)
- CKD3: with clinical symptoms and signs of kidney injury, and 30<=GFR<=59（ml/min/1.73m²)
- CKD4: with clinical symptoms and signs of kidney injury, and 15<=GFR<=29（ml/min/1.73m²)
- CKD5: with clinical symptoms and signs of kidney injury, and GFR<15（ml/min/1.73m²)

SUMMARY:
Patients with chronic renal insufficiency usually develop secondary osteoporosis or bone loss, which is called renal osteodystrophy. Most of the previous studies focused on bone metabolism of patients in late stage of chronic renal insufficiency, especially those with chronic dialysis. In this study, bone metabolism of patients in different stages of chronic renal insufficiency will be observed to reveal the mechanism of development of renal osteodystrophy and provide clues for early intervention on renal osteodystrophy.

DETAILED DESCRIPTION:
In this study, patients with chronic renal insufficiency (CKD1-5, defined by glomerular filtration rate，GFR) and healthy people as control will be recruited (50/group, total 300). Blood urea nitrogen, creatinine,lumbar and hip bone mineral density, bone turnover biochemical markers including serum total propeptide of type I procollagen（PINP）, bone alkaline phosphatase（BALP）, bone Gla-protein (BGP) and β-CrOSSlaps（β-CTX）, serum calcium and phosphorus and related regulators including fibroblast growth factor 23 (FGF23), 25-hydroxyl-Vitamin D （25-OH-VitD）, parathyroid hormone（PTH） will be detected. The relationship between kidney function and bone turnover, and the rules throughout the development process of renal osteodystrophy will be analysed.The micro ribonucleotide（miRNA）array will also be performed to screen the biomarkers of renal osteodystrophy in different stage.

ELIGIBILITY:
Inclusion Criteria:

1. 20-50 years old
2. chronic renal insufficiency (Control: normal kidney function; Case: CKD 1-5)
3. be willing to and be able to join in the study and signed informed consent
4. have not accepted systematical treatment on bone loss or osteoporosis

Exclusion Criteria:

1. allergies
2. secondary osteoporosis caused by other diseases.
3. postmenopausal women
4. mental illness or psychosis
5. patients with bone fracture and need surgery treatment
6. taking any medicine that will affect bone metabolism for a long time and can not stop
7. women during pregnant stage and breast-feed stage
8. with deformity or disability

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Cases groups (CKD-5) are recruited from inpatients and outpatients in the 4 centers.
  Controls are recruited from community samples and physical examination population.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-10 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
bone metabolism (bone mineral density and serum bone turnover biomarkers) | 1 day after enrollment
  lumbar (L1-4 as well as total) and hip (neck, troch, inter and word's) bone mineral density will be recorded by dual energy X-ray absorptiometry. Serum bone turnover biomarkers including total PINP, BGP, BALP and β-CTx will be detected.

SECONDARY OUTCOMES:
Kidney function （blood creatinine and urea nitrogen,glomerular filtration rate） | 1 day after enrollment
  CKD1-5 will be graded by glomerular filtration rate,and blood creatinine and urea nitrogen will be detected.
Calcium and phosphorus metabolism (serum calcium and phosphorus,calcium-phosphorus product, FGF23, PTH and 25-OH-VitD) | 1 day after enrollment
  Serum calcium and phosphorus will be detected and the calcium-phosphorus product will be calculated.Factors which are related with calcium and phosphorus including FGF23, PTH and 25-OH-VitD will be detected.
MicroRNA array | 1 day after enrollment
  Blood plasma will be collected for microRNA array analysis to find specific biomarkers for each stage.We will also try to find biomarkers for better definitions of chronic renal insufficiency and renal osteodystrophy.

OTHER OUTCOMES:
Baseline information （height, weight, sex） | 1 day after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun Wang, Doctor, Principal Investigator — Shanhgai University of TCM
Locations (4):
- China (4):
  - Anhui Province Hospital of TCM, Hefei, Anhui
  - Jiangsu Province Hospital of TCM, Nanjing, Jiangsu
  - Longhua hospital affiliated to Shanghai University of TCM, Shanghai, Shanghai Municipality
  - Huadong Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality